CLINICAL TRIAL: NCT06394024
Title: Examination of Postdural Puncture Headache Frequency, Predisposing Factors and Treatment Applied in Patients Undergoing Spinal Anesthesia
Brief Title: Examination of Postdural Puncture Headache Frequency, Predisposing Factors and Treatment
Acronym: PDPH
Status: Completed | Type: Observational
Sponsor: Mustafa Soner Ozcan (Other)
Responsible Party: Sponsor-Investigator, Mustafa Soner Ozcan, medical doctor, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Other Study IDs: İLK-10-124
Record Dates: First submitted 2024-04-16; First posted 2024-05-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- POSTDURAL PUNCTURE HEADHECHE: We don't use drug

SUMMARY:
Post-dural puncture headache (PDPH) is one of the most important complications of neuraxial blocks and lumbar interventions for cerebrospinal fluid (CSF) examination. It occurs due to tear in the dura mater and loss of cerebrospinal fluid (CSF) after intrathecal or epidural interventions.The incidence of PDPH depends on the thickness of the needle used and the type of tip. Headaches are more common with thick needles than with thin needles.In our study, postdural puncture headache in patients whose surgery was planned and spinal anesthesia was applied at Süleyman Demirel University faculty of medicine;frequency, predisposing factors, treatment intended to examine.

DETAILED DESCRIPTION:
Different anesthesia techniques are applied to patients undergoing surgery. These are general anesthesia and regional (Spinal, Epidural, peripheral nerve blocks, etc.) anesthesia applications. Today, regional anesthesia is the most frequently preferred anesthesia method by anesthesiologists due to its low side effects. Spinal anesthesia is the temporary stopping of nerve conduction with a local anesthetic solution injected into the cerebrospinal fluid. It is one of the most commonly used regional anesthesia techniques today.Important advantages of regional anesthesia include the patient's continued spontaneous breathing, preservation of oropharyngeal reflexes, continuation of analgesia in the postoperative period, early mobilization, and short hospital stay.Post-dural puncture headache (PDPH) is one of the most important complications of neuraxial blocks and lumbar interventions for cerebrospinal fluid (CSF) examination. The incidence of PDPH is significantly higher in young people than in the elderly, in women compared to men, and in pregnant women compared to the normal population.In our study, spinal anesthesia cases will be examined. Patients with headache will be identified. Patients' demographic data (age, height, body weight, gender, comorbidities), ASA (American Society of Anesthesiologists) score, operation type, presence of headache etiology, needle type and diameter used, number of interventions and procedures. level, amount of local anesthetic given, adjuvant drugs added, experience of the practitioner, amount of fluid given, date and time of headache onset, treatment and procedure complications will be monitored and recorded in the form.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* ASA physical status class I, II and III
* BMI <40 kg/m²
* Patients undergoing spinal anesthesia

Exclusion Criteria:

* ASA physical status class > III
* Severe cardiac, respiratory, hepatic, and renal disease
* Refusing spinal anesthesia
* History of local anesthetic allergy
* Localized infection at the injection site
* Coagulopathy
* Anticoagulant drugs usage
* History of chronic pain (migraine, sinusitis, etc.)
* Alcohol and opioid addiction
* Psychiatric diseases
* Communication difficulties
* Vertebral or chest wall abnormalities
* BMI > 40 kg/m²

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18 years and over
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
postdural puncture headache frequency | 6 months
  -rate of headache
postdural puncture headache treatments | 6 months
  -rate of treatments,
Number of patients receiving postdural puncture headache treatments | 6 months
  -number of participants
is postdural puncture headache treatments successful? | 6 months
  -success of treatment participants were also asked about the success of their treatment; the answer was yes or no.
number of patient having postdural puncture headache | 6 months
  -number of participants

SECONDARY OUTCOMES:
Relationship between postdural puncture headache and predisposing factors | 6 months
  -rate of headache
Number of patients obtained as a result of the relationship between postdural puncture headache and predisposing factors | 6 months
  -number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Soner Mustafa Soner, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No